CLINICAL TRIAL: NCT07197671
Title: Phase 1 Study of Y-NM600 in Patients Receiving Anti-PD-1 or Anti-PD-L1 Therapy for Metastatic Cancer
Brief Title: Y-NM600 in Patients Receiving Anti-PD-1 or Anti-PD-L1 for Metastatic Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Archeus Technologies, Inc. (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0647; SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); Protocol Version 10/31/25 (Other: UW Madison); UW24136 (Other: OnCore ID); P50CA278595-06A1 (NIH)
Record Dates: First submitted 2025-09-15; First posted 2025-09-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 3x3 dose escalation
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase 1A: Dose Level -1 (Experimental): 20 mCi x 1 90Y-NM600
  Interventions: Drug: 90Y-NM600
- Phase 1A: Dose Level 1 (Experimental): 35 mCi x 1 90Y-NM600
  Interventions: Drug: 90Y-NM600
- Phase 1A: Dose Level 2 (Experimental): 70 mCi x 1 90Y-NM600
  Interventions: Drug: 90Y-NM600
- Phase 1A: Dose Level 3 (Experimental): 105 mCi x 1 90Y-NM600
  Interventions: Drug: 90Y-NM600
- Phase 1A: Dose Level 4 (Experimental): 140 mCi x 1 90Y-NM600
  Interventions: Drug: 90Y-NM600
- Phase 1B: Single Dose (Experimental): Informed by Phase 1A
  Interventions: Drug: 90Y-NM600
- Phase 1B: Multi-dose (Experimental): Informed by Phase 1A and Single Dose Phase 1B
  Interventions: Drug: 90Y-NM600

INTERVENTIONS:
Drug: 90Y-NM600 — NM600 is a tumor-selective, pan-cancer, targeted radionuclide therapy (TRT) with theranostic capacity
  Other Names: alkylphosphocholine (APCh) analog

SUMMARY:
Participants with metastatic cancer who are taking anti-PD-1 or anti-PD-L1 therapy will be enrolled to assess the safety of and find the optimal dose for radioactive imaging agents and to explore whether these agents will make current drug therapies work better. Up to 60 participants will be enrolled and can expect to be on study for up to 9 months.

DETAILED DESCRIPTION:
This is a safety study of 86Y-NM600 and 90Y-NM600 and a dose finding study for 90Y-NM600 in patients with metastatic cancers who are receiving anti-PD-1 or anti-PD-L1 therapy and have immune-unconfirmed progressive disease (iUPD). The imaging agent 86Y-NM600 will be injected, and serial positron-emission tomography (PET)/computed tomography (CT) imaging will be performed to enable dosimetry calculations that will be used to determine eligibility for 90Y-NM600.

Phase 1a of the study (dose finding) will enroll 6-24 participants into a 3x3 dose finding plan where 3 participants start at Level 1 (below) and the number of participants with dose limiting toxicities (DLTs) will inform the next 3 participants:

* 0/3 Escalate to next higher dose level*
* 1/3 Accrue additional 3 patients at current dose level
* 1/3 + 0/3 Escalate to next higher dose level*
* 1/3 + ≥ 1/3 End phase 1a or de-escalate to dose level -1 if at dose level 1
* ≥ 2/3 End phase 1a or de-escalate to dose level -1 if at dose level 1

Dosing Plan:

* Level -1: 20 millicurie (mCi) x 1
* Level 1: 35 mCi x1
* Level 2: 70 mCi x1
* Level 3: 105 mCi x1
* Level 4: 140 mCi x1

Phase 1b (expansion cohort) may enroll up to an additional 36 participants (18 into a single dose cohort, 18 into a multi-dose cohort) with metastatic cancer.

The primary endpoints are to determine the safety of administering 86Y-NM600 for imaging and 90Y-NM600 for delivering radiation in patients with iUPD metastatic cancer who are receiving standard-of-care anti-PD-1 or anti-PD-L1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be informed of the investigational nature of the study and must be able to sign a written informed consent.
2. Participants with histologically or cytologically confirmed squamous cell carcinoma thought to originate from the head and neck region (HNC).
3. Participants must have metastatic disease of one of the following types: bile duct cancer, bladder cancer, cervical cancer, colorectal cancer, cutaneous squamous cell cancer, esophageal cancer, head and neck squamous cell carcinoma, kidney cancer, liver cancer, lung cancer, melanoma, merkel cell carcinoma, mesothelioma, stomach cancer, triple-negative breast cancer, or any solid cancer with mismatch repair deficiency.
4. Participants must be under treatment with one of the following standard-of-care anti-PD-1 or anti-PD-L1 therapies that is FDA approved for the patient's specific type of metastatic cancer: Pembrolizumab (Keytruda; anti-PD-1 antibody), Nivolumab (Opdivo; anti-PD-1 antibody), Atezolizumab (Tecentriq, anti-PD-L1 antibody), Avelumab (Bavencio; anti-PD-L1 antibody), Durvalumab (Imfinzi; anti-PD-L1 antibody), Cemiplimab (Libtayo; anti-PD-1 antibody), Dostarlimab (Jemperli; anti-PD-1 antibody). The patient must also have iUPD (Immune Unconfirmed Progressive Disease) after most recent imaging studies and be eligible to continue anti-PD-1 or anti-PD-L1 therapy, per the treating physician.

   1. For the purposes of this study, patients will be considered to have iUPD if they have been on treatment with anti-PD-1 or anti-PD-L1 therapy for any duration of time and, on their most recent standard-of-care imaging, been observed to have evidence of progression when the most recent scans prior to those did not show evidence of progression. Evidence of progression in this context will be defined as a 20 percent or greater increase in the sum of diameters of up to 5 lesions (these lesions will be identified as representative of the distribution of the patient's metastatic disease by the treating physician), the appearance of a new lesion, or the unequivocal progression of any lesion.
   2. Participants with iUPD standardly continue on anti-PD-1 or anti-PD-L1 therapy if the treating physician determines they do not have worsening performance status, clinically relevant increase in disease-related symptoms, or requirement of intensified management of disease-related symptoms. To be eligible for study, a participant's treating physician must determine that it is in the patient's best interest to continue on their current immune checkpoint inhibition regimen for additional treatment cycles until the subject's next scheduled standard-of-care imaging assessment. Treating physicians making this decision should generally do so if they feel the subject has no available better alternative treatment approach.
   3. In addition to anti-PD-1 or anti-PD-L1 therapy, patients may also be under treatment with and may continue to receive Ipilimumab (Yervoy; anti-CTLA4 antibody) or Tremelimumab (Imjuno; anti-CTLA4 antibody) during this study. However, participants must have been found to have iUPD while on the immune checkpoint therapy regimen that they receive during this study (i.e., participant's treating physician must determine that it is in the participant's best interest to stay on the current regimen of immune checkpoint inhibition until the subject's next standard of care imaging evaluation).
5. Participants must have received and shown evidence of progression or iUPD on at least one front-line therapy for metastatic disease. This can include the immune checkpoint inhibitor they are currently taking.
6. Participants must have at least one evaluable (measurable) tumor that is radiographically detectable.
7. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
8. Participants must have a life expectancy of at least 6 months.
9. People who could become pregnant have a confirmed negative urine pregnancy test within 7 days prior to receiving Y-NM600.
10. Participants must use a medically acceptable method of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence during the study participation and for 6 months after last dose of study drug. Participants who are postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) are not considered to be people who could become pregnant.
11. Participants who are not surgically or medically sterile agree to use an acceptable method of contraception. Participants who could impregnate their sexual partners must abstain from intercourse for three weeks after Y-NM600 treatment and agree to use condoms at least 2 months after the last dose of this drug. Total abstinence for the same study period is an acceptable alternative.
12. The participant has adequate renal function as defined by Cockcroft-Gault calculated creatinine clearance >60 ml/min
13. The subject has adequate hepatic function as defined by:

    1. total bilirubin ≤ 1.5 times the upper limit of normal (ULN)
    2. aspartate transaminase (AST) and alanine transaminase (ALT) less than or equal to 3.0 times the ULN
14. The participant has adequate hematologic function without Granulocyte-Macrophage Colony-Stimulating Factor (GM-CSF) injection or transfusion in the prior 7 days, as evidenced by:

    1. an absolute neutrophil count (ANC) greater than or equal to 2000 / μL
    2. hemoglobin greater than or equal to 8 g/dL
    3. platelets greater than or equal to 100,000 / μL, or, if full-dose anticoagulation therapy is used, platelets greater than or equal to 150,000 / μL are required.
    4. lymphocytes greater than or equal to 1000 / μL
15. For phase 1a, participant must be willing to undergo 2 core needle biopsies that are accessible via ultrasound and/or clinical biopsy.
16. Adequate uptake of 86Y-NM600 (3x red bone marrow) on PET CT imaging as determined by Nuclear Medicine.
17. No grade 2 toxicities new compared to baseline and unrelated or unlikely related to disease or any known cause other than 86Y-NM600 were noted through day 7 after 86Y-NM600 infusion.
18. No grade greater than or equal to 3 toxicities new compared to baseline were noted through day 7 after 86Y-NM600 infusion.

Exclusion Criteria:

1. Other concurrent severe and/or uncontrolled concomitant medical or psychiatric conditions (e.g., active or uncontrolled infection, uncontrolled diabetes) that could cause unacceptable safety risks or compromise compliance with the protocol, per investigator discretion.
2. The participant is taking strong inducers or inhibitors of CYP450 enzymes or drug transporters that cannot be held from at least 30 days prior to administration of 86Y-NM600 through the final 90Y-NM600 infusion without any expected adverse events. Examples include: clarithromycin, erythromycin, diltiazem, itraconazole, ketoconazole, ritonavir, verapamil, phenobarbital, phenytoin, rifampicin, and glucocorticoids.
3. Chemotherapy, radiotherapy, or major surgery within 3 weeks prior to study enrollment (this will be greater than 5 weeks prior to 90Y-NM600 therapy).

   a. For patients receiving prior radiation therapy, the dose to tumor, kidneys, liver, and bone marrow must be recorded, if available.
4. The participant is pregnant, breastfeeding, or expecting to conceive or could impregnate someone within the projected duration of the trial, starting with the screening visit through 6 months after the last dose of trial treatment.
5. Any ongoing or active infection, including active tuberculosis, hepatitis B or C, or known infection with the human immunodeficiency virus (HIV) that is not well controlled (undetectable viral load by PCR) by anti-retroviral therapy.
6. Concurrent treatment with any other systemic anti-cancer or investigational agents other than an anti-PD-1, anti-PD-L1, or anti-CTLA-4 antibody. Subjects cannot be receiving concomitant chemotherapy, experimental therapy or any other therapy not otherwise outlined by the trial for the purposes of anti-cancer treatment.

   b. Palliative external beam radiation therapy may be delivered to patients during this study if deemed necessary and safe by the treating physician.

   c. Participants can be receiving dual immune checkpoint inhibition with an anti-CTLA-4 antibody in addition to an anti-PD-1 or anti-PD-L1 therapy.
7. Patients with a history of or concurrent second primary malignancy within 2 years to study enrollment are excluded, with the exception of patients who have had definitive treatment of a primary skin basal cell, skin squamous cell carcinomas, or localized low or intermediate risk prostate cancer - these subjects are eligible 3 months after completion of definitive treatment for that prior cancer.
8. Participants that have had total body or hemibody irradiation, or have had prior systemic radioisotope therapy (except for benign thyroid disease)
9. Any condition requiring the use of immunosuppression, excluding rheumatologic conditions or endocrine conditions treated with stable doses of corticosteroids (equivalent to prednisone 10 mg daily)
10. Ongoing hemodialysis or peritoneal dialysis
11. Any known medical condition that predisposes the subject to uncontrolled bleeding such as hemophilia or clotting factor deficiencies
12. Participants with known genetic conditions causing pre-disposition to RT toxicity (i.e.: Li-Fraumeni, ataxia telangiectasia mutated (ATM) deficiency, active scleroderma, active inflammatory bowel disease, active systemic lupus)
13. Patients with an implanted defibrillator or with an implanted pacemaker and pacemaker dependency for rate or rhythm control
14. Patients with repeated demonstration on two EKGs of a QTcF interval greater than 470 milliseconds or use of medications known to prolong the QT/QTc interval
15. Participants who cannot provide independent, legal, informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Toxicities greater than or equal to Grade 3 at least possibly related to 86Y-NM600 | baseline screening, Day 7 after 86Y-NM600 injection
  Toxicities greater than or equal to Grade 3 at least possibly related to 86Y-NM600 by day 7 (greater than 10 half-lives of 86Y) after 86Y-NM600 injection, as defined by the NCI CTCAE version 5.0.
Toxicities greater than or equal to Grade 3 at least possibly related to 90Y-NM600 | up to 9 months on study
  Toxicities greater than or equal to Grade 3 at least possibly related to 90Y-NM600 by day 42 after final 90Y-NM600 injection, as defined by the NCI CTCAE version 5.0.
  Time points of investigation include:
  * baseline screening
  * Phase 1A: post injection week 1, week 2, week 3, week 4
  * Phase 1B: 7 days after each injection, 30 days and 42 days after final injection

SECONDARY OUTCOMES:
Pharmacokinetics of Y-NM600: Blood concentration verse time curve | 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hour, and *48 hours after infusion (*Phase 1A only)
  Blood concentration verse time curve, blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hour, and *48 hours after infusion (*Phase 1A only)
Pharmacokinetics of Y-NM600: Time to reach maximum concentration of Y-NM600 in Blood | Blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hour, and *48 hours after infusion (*Phase 1A only)
  Blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hour, and *48 hours after infusion (*Phase 1A only)
Pharmacokinetics of Y-NM600: Blood Radioactivity from Y-NM600 | Blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hours, and *48 hours after infusion (*Phase 1A only)
  Blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hour, and *48 hours after infusion (*Phase 1A only)
Pharmacokinetics of Y-NM600: Physiological Half-life of Y-NM600 | Blood draws at estimated Cmax 3-5 min after end of infusion, 0.5 hours, *2.0 hours, 4.0 hours, 24 hours, and *48 hours after infusion (*Phase 1A only)
  Phase 1a: Blood draws at estimated Cmax 3-5 min after end of infusion (+/- 5 min), 0.5 hours (+/- 15 min), 2.0 hours (+/- 30 min), 4.0 hours (+/- 30 min), 24 hours (+/- 120 min), and 48 hours (+/- 120 min) after infusion.
  Phase 1b: Blood draws at estimated Cmax 3-5 min after end of infusion (+/- 5 min), 0.5 hours (+/- 15 min), 4.0 hours (+/- 30 min), and 24 hours (+/- 120 min) after infusion.
  Cumulative urine collection will be done for 6 hours with specific samples collected and pooled at 0.5 hours (+/- 15 min), 3 hours (+/- 30 min), and at 5 hours (+/- 30 min) after infusion.
Proportion of Participants with 3-fold or greater uptake of 86Y-NM600 in tumor site compared to red bone marrow | 48-72 hours after 86Y-NM600 infusion
  Assessed via PET/CT 48-72 hours after 86Y-NM600 infusion as Maximum Standardized Uptake Value (SUVmax) at tumor sites previously identified by standard of care imaging and at a site of red bone marrow.
Overall Response Rate (ORR) by iRECIST at 8 weeks after initial 90Y-NM600 injection (D1) | baseline, standard-of-care imaging 8 weeks after D1
  ORR will include iCR and iPR and will be determined as per iRECIST, by investigator assessment.
Safe and Effective Dose Level for Phase 1B | Phase 1A: baseline, Once per week for four weeks after 90Y-NM600 injection and at day 42 after 90Y-NM600 injection, Standard-of-care imaging 8 weeks after D1 of 90Y-NM600
  A recommended phase 1b single treatment dose level is based on the following criteria: 1) a dose level resulting in less than 33 percent of participants with Dose Limiting Toxicities by 42 days after final 90Y-NM600 injection, 2) the dose level with the greatest ORR among dose levels that meet criteria 1 and the lower dose level if ORR is equal at two dose levels, and 3) the highest dose level that meets criteria 1 if no participants exhibit ORR in any regimen that meets criterion 1.
  For the multi-dose expansion cohort, the recommended dose will be the single treatment expansion dose level or the next highest dose level for which OLINDA calculations from PET/CT imaging at 48-72 hours after 86Y-NM600 for all enrolled patients predict cumulative mean doses of less than 23 Gy to the kidney, less than 2 Gy to the red bone marrow, and less than 30 Gy to liver in greater 66 percent of participants following three cycles of 90Y-NM600 at the multi-dose expansion cohort dose level.

OTHER OUTCOMES:
Progression Free Survival (PFS) | Day 1 of treatment, Standard-of-care imaging follow-up ~3 and 6 months after Day 1, Time of disease progression (monitored up to 5 years)
  PFS is defined as the time from Day 1 of treatment until the criteria for disease progression is met as defined by iRECIST or death as a result of any cause.
Overall Survival (OS) | Day 1 of treatment, Standard-of-care imaging follow-up ~3 and 6 months after Day 1, Time of disease progression, Death (monitored up to 5 years)
  OS is defined as time from Day 1 of treatment until death as a result of any cause.
Duration of Response | Day 1 of treatment, Standard-of-care imaging follow-up ~3 and 6 months after Day 1, Time of disease progression (monitored up to 5 years)
  Duration of response is the period measured from the time that measurement criteria are met for immune complete response (iCR), immune partial response (iPR), or immune-related stable disease (iSD) (whichever status is recorded first) until the date that recurrent or iPD is objectively documented.
EORTC QLQ-C30 | baseline, 1 week after Day 1, 8 weeks after Day 1
  Determine the impact of 90Y-NM600 on patient-reported health-related quality of life (HRQoL) by assessing the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30). The EORTC QLQ-C30 is scored from 0-100 where higher scores indicate a better quality of life.
EQ-5D Score | baseline, 1 week after Day 1, 8 weeks after Day 1
  Determine the impact of 90Y-NM600 on patient-reported health-related quality of life (HRQoL) by assessing the EQ-5D. The EQ-5D is scored between 0-1 where better quality of life is closer to 1.
Tumor Heterogeneity | PET/CT imaging at 1-6 hours, 18-36 hours, and 48-72 hours after 86Y-NM600 infusion
  Mean, minimum, and maximum dose predicted for 86Y-NM600 and 90Y-NM600 in tumors greater than 2 cm and for select normal organs [kidney, liver, red bone marrow, blood (2 cm region of abdominal aorta that is great than 1 cm away from any identified tumor site)] will be determined from three serial 86Y-NM600 PET/CT images. When feasible, this will be performed for all tumor sites greater than 2 cm in any diameter. If the reading radiologist determines this is not feasible, then 5 tumors greater than 2cm will be randomly chosen and dosimetry evaluated at these sites.
Tumor Expression of Immune Susceptibility Markers | Pre-treatment baseline, 1 week after Day 1
  Expression of PD-L1, MHC-1, VCAM-1, and IFNβ mRNA by polymerase chain reaction (PCR) on CD45- cells isolated from disaggregated tumor biopsies.
90Y-NM600 Tumor Microenvironment Immunologic Activation | Pre-treatment baseline, 1 week after Day 1
  Sorted CD45+ cells isolated from disaggregated tumor biopsies will be analyzed by scRNAseq
Count of Circulating Tumor Cells (CTCs) | Pre-treatment baseline, 1 week after Day 1
  CTCs captured by CapioCyte will be quantified, radioactivity directly measured, and mRNA extracted for PCR analysis of PD-L1, MHC-1, VCAM-1, and IFNβ expression.
Radioactivity of Circulating Tumor Cells (CTCs) | Pre-treatment baseline, 1 week after Day 1
  CTCs captured by CapioCyte will be quantified, radioactivity directly measured, and mRNA extracted for PCR analysis of PD-L1, MHC-1, VCAM-1, and IFNβ expression.
Expression of Circulating Tumor Cells (CTCs) | Pre-treatment baseline, 1 week after Day 1
  CTCs captured by CapioCyte will be quantified, radioactivity directly measured, and mRNA extracted for PCR analysis of PD-L1, MHC-1, VCAM-1, and IFNβ expression.
Phenotype of CD8+ T cells | Pre-treatment, Every 4 weeks after Day 1
  Peripheral blood mononuclear cells (PBMCs) will be sorted to isolate CD8+ T cells and these will be evaluated by IsoPlexis single cell proteomics assay and by deep sequencing of the T cell receptor.
Mutation Burden of Circulating Tumor DNA | Pre-treatment baseline, 1 week after Day 1
  Measure changes in ctDNA fraction, tumor mutation burden, and the clonal evolution of tumors with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Blitzer, MD, Principal Investigator — UW Carbone Cancer Center; Justine Bruce, MD, Principal Investigator — UW Carbone Cancer Center; Zachary Morris, PhD, Study Chair — UW Carbone Cancer Center; Paul Harari, MD, Study Chair — UW Carbone Cancer Center
Locations (1):
- UW Carbone Cancer Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF